CLINICAL TRIAL: NCT00632710
Title: Assessment of the Effectiveness of Low-Level Laser Therapy on the Hands of Patients With Rheumatoid Arthritis: a Randomized Double-Blind Controlled Trial
Brief Title: Assessment of the Effectiveness of Low-Level Laser Therapy on the Hands of Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Rheumatology Division, Federal University of Sao Paolo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0829/04; FAPESP 2004/09374-1; CNPQ grant
Record Dates: First submitted 2008-02-07; First posted 2008-03-11 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; hands; randomized controlled; low level laser
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- b (Experimental): laser
  Interventions: Other: phototherapy
- a (Placebo Comparator): laser placebo
  Interventions: Other: phototherapy placebo

INTERVENTIONS:
Other: phototherapy — The laser used was low-level Aluminum Gallium Arsenide (AlGaAs)diodo laser, at a wavelength of 785 nm (infrared), dose of 3 J/cm2, mean power of 70 mW, 3 sec. per point, laser beam of 0,06cm2, BIOSET brand - Indústria de Tecnologia Eletrônica Ltda -Rio Claro, Brazil.
  Other Names: soft laser therapy
  Arms: b
Other: phototherapy placebo — disconnected laser (same device - experimental group)
  Other Names: soft laser placebo therapy
  Arms: a

SUMMARY:
The purpose of the present study was to assess the effectiveness of low-level laser therapy on the reduction in pain and improvement in function in the hands of patients with rheumatoid arthritis

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease of unknown etiology that basically compromises the joints in a generalized, symmetrical, additive and usually progressive manner. This clinical condition includes pain and altered functionality. Low-level laser therapy (LLLT) has been studied since the 1970s with regard to its therapeutic effects. The literature suggests that it offers analgesic as well as anti-inflammatory benefits.

A number of studies carried out in the laboratory and on animals have shown that LLLT contributes toward the treatment of inflammatory joint disease. However, studies on humans with RA have yielded controversial results. A large part of the authors researched state that further randomized double-blind controlled studies should be carried out to prove the effectiveness of LLLT on RA. Thus, the aim of the present study was to assess the effectiveness of LLLT on the reduction in pain and improvement in function in the hands of patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* patients with RA
* inflammatory condition of at least two hand joints among the wrists, proximal interphalangeal (PIP) joint and metacarpophalangeal (MCP) joint
* visual analogue scale (VAS) for pain between 3 and 8 cm during activities of daily living
* and being of either gender

Exclusion Criteria:

* skin lesions at the application site
* other illnesses affecting the hands; physiotherapy for the hands in the previous three months
* joint injections in the previous three months
* change in disease-modifying anti-rheumatic drugs in the previous three months
* and change in corticosteroids in the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
pain | 2 months

SECONDARY OUTCOMES:
function | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Meireles, Physiother., Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Federal University of Sao Paulo — http://www.unifesp.br
- See also: Brazilian Coordination of Upper Education Personal Improvement — http://www.capes.gov.br
- See also: Sao Paulo State Research Assistance Foundation — http://www.fapesp.br